CLINICAL TRIAL: NCT01438762
Title: Early Intervention for Adolescents With Patellofemoral Pain Syndrome - a Cluster Randomized Trial
Brief Title: Early Intervention for Adolescents With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mogens Berg Laursen (Other)
Collaborators: University of Southern Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Mogens Berg Laursen, Administrator, Northern Orthopaedic Division, Denmark
Organization: Northern Orthopaedic Division, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20110020
Record Dates: First submitted 2011-08-02; First posted 2011-09-22 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Anterior Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Educational Status; Standard of Care; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Information and patient education (Active Comparator): All subjects will receive one-to-one patient education delivered by a physiotherapist. The information will be standardized and cover the topics of: why does it hurt: pain management; information of how to reduce physical activity if necessary; how to return slowly to sports; how to cope with knee pain and information of how to increase knee alignment during walking and stair walking. The patients will also receive this information in written form. This information is expected to take approximately 45minutes per patient.
  Interventions: Behavioral: Patient information and education
- Information, education and physiotherapy (Active Comparator): Patients will receive one-to-one patient education delivered by a physiotherapist. The information will be standardized and cover the topics of: why does it hurt: pain management; information of how to reduce physical activity if necessary; how to return slowly to sports; how to cope with knee pain and information of how to increase knee alignment during walking and stair walking.
  In addition the patients will receive supervised multimodal physiotherapy carried out by a physiotherapist with previous experience in treating adolescents and PFPS and has more than two years of practical experience in these areas.
  Interventions: Other: Information, education and physiotherapy
- Observational cohort (No Intervention): Those who do not wish to participate in the randomization procedure will be followed through an observational cohort. The observational cohort will be followed at the same time-points and they will be asked which treatment they have received.

INTERVENTIONS:
Behavioral: Patient information and education — All subjects will receive one-to-one patient education delivered by a physiotherapist. The information will be standardized and cover the topics of: why does it hurt: pain management; information of how to reduce physical activity if necessary; how to return slowly to sports; how to cope with knee pain and information of how to increase knee alignment during walking and stair walking. The patients will also receive this information in written form. This information is expected to take approximately 45minutes per patient.
  Other Names: Standard care
  Arms: Information and patient education
Other: Information, education and physiotherapy — Patients will receive one-to-one patient education delivered by a physiotherapist. The information will be standardized and cover the topics of: why does it hurt: pain management; information of how to reduce physical activity if necessary; how to return slowly to sports; how to cope with knee pain and information of how to increase knee alignment during walking and stair walking. The patients will also receive this information in written form.
  In addition the patients will receive supervised multimodal physiotherapy carried out by a physiotherapist with previous experience in treating adolescents and PFPS and has more than two years of practical experience in these areas. The multimodal physiotherapy intervention will be carried out at school premises right after the end of class.
  Other Names: Physiotherapy; Multimodal intervention
  Arms: Information, education and physiotherapy

SUMMARY:
Self-reported, unspecific knee pain is highly prevalent among adolescents. A large proportion of the unspecific knee pain can be attributed to Patellofemoral Pain Syndrome (PFPS). There are a number of treatment options for PFPS. Physical therapy has been advocated as one of the cornerstones in rehabilitation of patients with PFPS. Twenty-five years ago, McConnell proposed a multimodal approach that combined several treatment options. The regimen included retraining of the vastus medialis oblique muscle through functional weight bearing activities. This exercise is combined with patellar taping, patellar mobilization, and stretching to improve patellar tracking, reduce pain, and enhance vastus medialis oblique muscle activation. Short term results (<12 months) indicates that multimodal physiotherapy is more effective than placebo treatment.

While treatment for PFPS may be successful for the short-term, long-term results are less promising. A recent review covering the long term prognosis for patients diagnosed with PFPS, reported that only 1/3 of those diagnosed with PFPS and treated conservatively were pain free 12 months after diagnosis. Further ¼ stopped participating in sports because of knee pain.

Predictors of long term outcome (>52weeks) indicate that a long symptom duration, higher age and greater severity at baseline are associated to poorer outcome after treatment. These prognostic factors suggest that an early initiation of treatment might lead to a better long-term prognosis. The purpose of this study is to examine the short and long-term effectiveness of multi-modal physiotherapy compared to standard wait-and-see treatment applied at a very early state of disease among adolescents. The investigators hypothesized a significantly larger proportion of completely recovered patients at three-month follow-up in the interventions group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-19 years
* Insidious onset of anterior knee or retropatellar pain of greater than six weeks' duration
* Provoked by at least two of prolonged sitting or kneeling, squatting, running, hopping, or stair walking
* Tenderness on palpation of the patella, or pain with step down or double leg squat
* Worst pain over the previous week of at least 30 mm on a 100 mm visual analogue scale.

Exclusion criteria:

* Concomitant injury or pain from the hip, lumbar spine, or other knee structures
* Previous knee surgery
* Patellofemoral instability
* Knee joint effusion
* Use of physiotherapy for treating knee pain within the previous year
* Use of weekly use anti-inflammatory drugs.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2011-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in perception of recovery after 12 months measured on a 7-point likert scale ranging from "completely recovered" to "worse than ever". | Baseline, 3, 6, 12 and 24months
  Perception of recovery after 12 months measured on a 7-point likert scale ranging from "completely recovered" to "worse than ever".

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | Baseline, 3, 6, 12 and 24months
EQ5D | Baseline, 3, 6, 12 and 24months
Neuromuscular function | Baseline and 3 months
  Each subjects will undergo quadriceps strength measurements and two basic tests of neuromuscular function of m. vastus medialis and m. vastus lateralis. EMG will be collected during two different conditions: Walking and semi-squat at 90 degrees flexion at the knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Rathleff, Principal Investigator — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Ewa M Roos, Ph.d, Study Chair — Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Denmark; Jens L Olesen, MD, Ph.d, Study Chair — Aalborg University Hospital; Sten Rasmussen, MD, Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark
Locations (1):
- Orthopaedic Surgery Research Unit, Aalborg Hospital, Aalborg, Aalborg, Denmark

REFERENCES:
- [Derived] Rathleff MS, Roos EM, Olesen JL, Rasmussen S. Exercise during school hours when added to patient education improves outcome for 2 years in adolescent patellofemoral pain: a cluster randomised trial. Br J Sports Med. 2015 Mar;49(6):406-12. doi: 10.1136/bjsports-2014-093929. Epub 2014 Nov 11. PMID 25388552
- [Derived] Rathleff MS, Roos EM, Olesen JL, Rasmussen S, Arendt-Nielsen L. Lower mechanical pressure pain thresholds in female adolescents with patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2013 Jun;43(6):414-21. doi: 10.2519/jospt.2013.4383. Epub 2013 Mar 18. PMID 23508216
- [Derived] Rathleff MS, Roos EM, Olesen JL, Rasmussen S. Early intervention for adolescents with patellofemoral pain syndrome--a pragmatic cluster randomised controlled trial. BMC Musculoskelet Disord. 2012 Jan 27;13:9. doi: 10.1186/1471-2474-13-9. PMID 22280484